CLINICAL TRIAL: NCT06005376
Title: Development of a Celiac Safe Food Additive: An Intervention Study in Healthy Volunteers
Brief Title: Development of a Celiac Safe Food Additive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Gothia Forum - Center for Clinical Trial (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Nathalie Scheers, Associate professor, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019F004
Record Dates: First submitted 2023-08-08; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Gluten Intolerance
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: Randomised double-blind crossover intervention
Who Masked: Participant, Care Provider
Masking Description: The participants did not know which bread was received; the bags were color-coded. The personnel meeting the participants did not know which color belonged to which bread. Only the principal investigator (and the bakery) not meeting participants knew which color belonged to which bread type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No additive (Active Comparator): This arm was served 2 reference wheat bread rolls (a 40 g) a day.
  Interventions: Other: Breakfast rolls consisting of wheat flour with and without a E304i/zinc additive
- E304i/zinc additive (Experimental): This arm was served 2 wheat bread rolls (a 40 g) a day containing a E304i/zinc additive.
  Interventions: Other: Breakfast rolls consisting of wheat flour with and without a E304i/zinc additive

INTERVENTIONS:
Other: Breakfast rolls consisting of wheat flour with and without a E304i/zinc additive — The participants were provided with two Breakfast rolls (a 40 g) a day during the intervention week. In addition, they were provided with gluten-free foods during the whole trial.

SUMMARY:
The goal of this clinical trial was to investigate if intestinal deamidation of gliadin from wheat bread could be hindered by adding a E304i/zinc additive. The study was a randomized double-blind 4-week crossover intervention in 20 healthy volunteers in which the participants ingested 2 bread rolls a day during the intervention weeks.

The question it aimed to answer was if there was a difference in blood levels of deamidated gliadin peptides after ingestion of the reference wheat bread compared with the wheat bread containing the food additive.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index between 18.5 to 32
* Age between 18-50 years
* No tobacco use

Exclusion Criteria:

* Celiac disease and other diagnosed enteropathies
* Gluten-free diet
* Dietary supplementation (minerals (calcium, zinc, vitamin D) and proteolytic enzymes, probiotics)
* Pregnancy or lactation
* Lack of suitability for participation in the study, for any reason, as judged by the medical doctor or the project PI.
* Withdrawn consent: Participant withdraws consent.
* Non-compliance: Participant fails repeatedly to comply with study protocol (diet, study visits and provide samples)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Levels of deamidated gliadin peptides in blood | Blood samples were drawn once weekly at day 7, 14, 21, 28
  Deamidated gliadin peptides in blood measured by ELISA using an antibody towards deamidated gliadin peptides

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Scheers, Principal Investigator — Chalmers University of Technology, Dept of Life Sciences, Gothenburg 412 96, Sweden
Locations (1):
- Chalmers University of Technology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The data and the study protocol will be published in a scientific journal. Participant data are anonymized and cannot be connected to an individual person.
Supporting Information: Study Protocol
Time Frame: As soon as published, no time limit
Access Criteria: The study will be published in an open access journal

REFERENCES:
- [Derived] Engstrom N, Bohn L, Josefsson A, Storsrud S, Scheers N. Development of celiac-safe foods: prevention of transglutaminase 2 (TG2) deamidation of gluten in healthy non-celiac volunteers. Front Nutr. 2024 Mar 14;11:1308463. doi: 10.3389/fnut.2024.1308463. eCollection 2024. PMID 38549745